CLINICAL TRIAL: NCT04554342
Title: Testing of a Candy in Five Different Versions for the Additional Humidification of the Oral Cavity (DESERTO)
Brief Title: Testing of a Candy in Five Different Versions for the Additional Humidification of the Oral Cavity
Acronym: DESERTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-01942; ex19Filippi3
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Xerostomia; Dryness of Mouth
Keywords: salivary flow rate; salivary flow stimulation
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: doppel- blind testing of 5 different variations of a candy in each participant by (unstimulated and stimulated) salivary flow rate; each participant is testing each variation of candy once in a randomized order at 5 consecutive days
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- healthy participants starting with candy V01 (Experimental): healthy participants testing a candy in 5 different variations by (unstimulated and stimulated) salivary flow rate (before and after comparison)
  Interventions: Other: V01 candy; Other: V02 candy; Other: V03 candy; Other: V04 candy; Other: V05 candy
- healthy participants starting with candy V02 (Experimental)
  Interventions: Other: V01 candy; Other: V02 candy; Other: V03 candy; Other: V04 candy; Other: V05 candy
- healthy participants starting with candy V03 (Experimental)
  Interventions: Other: V01 candy; Other: V02 candy; Other: V03 candy; Other: V04 candy; Other: V05 candy
- healthy participants starting with candy V04 (Experimental)
  Interventions: Other: V01 candy; Other: V02 candy; Other: V03 candy; Other: V04 candy; Other: V05 candy
- healthy participants starting with candy V05 (Experimental)
  Interventions: Other: V01 candy; Other: V02 candy; Other: V03 candy; Other: V04 candy; Other: V05 candy

INTERVENTIONS:
Other: V01 candy — candy with sweetener (Isomalt) and apple flavour
Other: V02 candy — candy with with sweetener (Isomalt) and apple flavour and acidifying agent (apple acid + citric acid)
Other: V03 candy — candy with with sweetener (Isomalt) and apple flavour and acidifying agent (apple acid + citric acid) and Vitamin C
Other: V04 candy — candy with sweetener (Isomalt) (control group 1)
Other: V05 candy — candy with with sweetener (Isomalt) and acidifying agent (apple acid + citric acid) (control group 2)

SUMMARY:
This study is to investigate whether a candy can increase moisture of the oral cavity and reduce dryness of mouth.

DETAILED DESCRIPTION:
A candy (available on the market from a Swiss manufacturer (Ricola)), free of ingredients that could interfere with the investigation, is tested in five different versions on different days. It is to analyse whether these candies can increase moisture of the oral cavity and reduce dryness of mouth.

ELIGIBILITY:
Inclusion Criteria:

* non- smoker
* no allergies
* no drug- use (except for contraception)
* healthy volunteers (no disease/infection 4 weeks before study participation)

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
dryness of mouth- sensation | one point assessment following consumption of candy (approx 5 minutes)
  dryness of mouth- sensation by Visual analogue scale (VAS); 0 = does not apply; 10 = is absolutely true.
Change in salivary flow rate (ml/min) | before and after consumption of candy (approx 5 minutes for each salivary flow measurement)
  Change in salivary flow rate (ml/min) before and after stimulation (mechanical and gustatory) by consumption of candy

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Filippi, Prof. Dr. med. dent., Principal Investigator — Universitäres Zentrum für Zahnmedizin Basel
Locations (1):
- Universitäres Zentrum für Zahnmedizin Basel, Basel, Switzerland